CLINICAL TRIAL: NCT00777686
Title: Quantifying Progression of Non-Enhancing Tumor in Patients With Recurrent Glioblastoma Treated With Antiangiogenic Agents
Brief Title: Measuring Non-Enhancing Glioblastoma Progression
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0492
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Brain Tumor; Glioblastoma
Keywords: Intracranial Glioblastoma; Intracranial Gliosarcoma; glioblastoma; recurrent glioblastoma; gliosarcoma; brain cancer; magnetic resonance spectroscopy; MRS; magnetic resonance imaging; MRI; MRI/MRS; Recurrent Glioblastoma Treated with Antiangiogenic agents; contrast enhanced MRI; DCE-MRI; diffusion-weighted MRI; DSC; DW-MRI
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Gliosarcoma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MRI/MRS Scanning: Magnetic resonance imaging with magnetic resonance spectroscopy (MRI/MRS Scanning)
  Interventions: Procedure: MRI/MRS Scan

INTERVENTIONS:
Procedure: MRI/MRS Scan — MRI/MRS brain scan with intravenous contrast prior to chemotherapy, then repeated every 8 weeks.
  Other Names: magnetic resonance spectroscopy; MR Imaging; MR; MRI/MRS scanning; MRI/MRS; MRI; MRS

SUMMARY:
The goal of this clinical research study is to learn if magnetic resonance imaging with magnetic resonance spectroscopy ("MRI/MRS" scanning) can measure any extra growth in the tumor that does not show up on regular MRI images. This study procedure will be performed on patients with recurrent glioblastoma who are either being treated with chemotherapy that blocks blood vessel growth, or will soon begin this type of chemotherapy.

DETAILED DESCRIPTION:
The Study Procedures:

MRI scanning is commonly used to check the status of glioblastoma. In this study, MRI scanning will also be used to try to better understand how chemotherapy that blocks blood vessel growth may be affecting the status of the glioblastoma.

The timing of all MRI scans for this study will be done on schedule for routine patient care. There will not be any extra MRI scans performed, but an MRS portion to the MRI scans will be added. The MRS results will be used in this study to look at the chemical differences between the cancerous and normal tissue, in order to try to better understand how your chemotherapy may be working.

Screening Tests:

Before you can begin this study, you will have "screening tests" to help the doctor decide if you are eligible to take part in this study. The following tests and procedures will be performed:

* Blood (about 1 teaspoon) will be drawn for routine tests.
* Women who are able to have children must have a negative blood (about 1 teaspoon) pregnancy test.

MRI/MRS Scanning:

If you are found to be eligible to take part in this study, you will have an MRI/MRS scan of the brain. The first of these scans will be performed before the chemotherapy starts (either before your first cycle of this type of chemotherapy or before your next cycle, depending on whether you were receiving this type of chemotherapy before the study or not). After that, an MRI/MRS scan will be repeated at Weeks 8 and 16 after the beginning of chemotherapy.

The MRI/MRS scans will follow the same procedure and use the same MRI scanner machine as a regular MRI scan, but will take about an additional 10 minutes. You will lie still on your back with your head placed within the openings of the scanner. A contrast solution, which helps make the tumor visible, will be given through a needle in your vein. The scanning procedure should take about an hour at each visit.

The results of the MRI/MRS scans will not be used to affect your course of treatment.

Tissue Collection:

If your regular doctor recommends that the tumor be surgically removed, the surgery will be discussed with you in detail and you will sign a separate informed consent form for it. Leftover tissue that was removed during the surgery will be collected and used as part of this study. The tissue will be used to further check the status of the disease, and it will be compared with the MRI/MRS images.

Biomarker Testing:

In this study, you will also have blood drawn for biomarker testing. Biomarkers are chemical "markers" in the blood, other body fluids, or tissue that may be related to the status of disease and/or the effects of treatment. This blood (about 2 teaspoons each time) will be drawn before the chemotherapy starts and then every 8 weeks while you are on study. The blood draws will occur on the same days as the MRI/MRS scanning.

Length of Study Participation:

You will continue having blood drawn for biomarker testing every 8 weeks, unless you stop taking this type of chemotherapy that blocks blood vessel growth. In that case, you will be taken off study.

If you do have surgery, your participation in this study will end after the surgery. If you are unable to have surgery, your participation will end after your last MRI/MRS scan.

This is an investigational study. MRI scanning is an FDA approved and commercially available procedure for checking the status of glioblastoma. At this time and for this purpose, MRS scanning is being used in research only.

Up to 18 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven intracranial glioblastoma or gliosarcoma will be eligible for this protocol
2. Patients with recurrent glioblastoma or gliosarcoma who are scheduled to start systemic chemotherapy with bevacizumab.
3. Patients tumor must be located in an area that is amenable to the proposed imaging sequences.
4. Patients must be age 18 or older.
5. Karnofsky Performance Status Scale (KPS) >/= 70.
6. Inclusion of Women and Minorities: Both men and women and members of all races and ethnic groups are eligible for this trial.
7. Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policies of the hospital. The only acceptable consent form is the one attached at the end of this protocol.

Exclusion Criteria:

1. Patients with histologically proven intracranial glioblastoma or gliosarcoma will be eligible for this protocol
2. Patients with recurrent glioblastoma or gliosarcoma who are scheduled to start systemic chemotherapy with bevacizumab.
3. Patients tumor must be located in an area that is amenable to the proposed imaging sequences.
4. Patients must be age 18 or older.
5. KPS >/= 70.
6. Inclusion of Women and Minorities: Both men and women and members of all races and ethnic groups are eligible for this trial.
7. Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policies of the hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, 18 years or older, with "recurrent" intracranial glioblastoma or gliosarcoma being treated with chemotherapy or will be treated.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2008-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Functional MR Measurements | Baseline, Every 8 weeks and at Off Study

CONTACTS AND LOCATIONS:
Overall Officials: John DeGroot, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org